CLINICAL TRIAL: NCT07303244
Title: The Association Between Eating and Sleep Attitudes and Perceived Stress as Predictors of Cardiovascular Risk Among Physical Therapy Students
Brief Title: Eating and Sleep Attitudes, Stress, and Cardiovascular Risk in Physical Therapy Students
Acronym: ESAS-CVR
Status: Enrolling by invitation | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Eldaly, Researcher, Cairo University
Other Study IDs: EGPHYSIO-SC-002
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Eating Attitudes; Lifestyle Risk Reduction; Perceived Stress
Keywords: Eating Attitudes; Cardiovascular Risk; Sleep Quality; Lifestyle Behaviors; Health Risk Prediction; Psychological Factors
MeSH Terms: conditions — Risk Reduction Behavior; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: complete validated questionnaires — Participants will only complete validated questionnaires (EAT-26, PSQI, PSS-10). No therapeutic or behavioral intervention will be administered.

SUMMARY:
The goal of this observational study is to assess how eating attitudes, sleep attitudes, and perceived stress contribute to early indicators of cardiovascular risk among undergraduate physical therapy students aged 18-30. The main questions it aims to answer are:

Do unhealthy eating attitudes correlate with increased perceived stress levels? Does poor sleep quality predict higher behavioral risk for cardiovascular disease?

Participants will complete validated self-reported questionnaires, including:

The Eating Attitudes Test (EAT-26) The Pittsburgh Sleep Quality Index (PSQI) The Perceived Stress Scale (PSS-10)

Data will be collected once, either electronically or on paper, and all responses will be coded anonymously. There is no intervention or comparison group, as the study is purely observational.

DETAILED DESCRIPTION:
This observational study explores how lifestyle-related psychological factors-including eating attitudes, sleep attitudes, and perceived stress-interrelate and contribute to early behavioral indicators of cardiovascular risk among undergraduate physical therapy students. The study focuses on a population frequently exposed to academic pressure, irregular schedules, and altered lifestyle habits, which may predispose them to long-term health risks.

Participants will complete three standardized self-report instruments: the Eating Attitudes Test (EAT-26), the Pittsburgh Sleep Quality Index (PSQI), and the Perceived Stress Scale (PSS-10). These tools were selected for their established validity in assessing eating behaviors, sleep quality, and stress perception in young adult populations. Scores from each measure will be analyzed to determine correlations among the variables and their combined ability to predict early cardiovascular risk patterns.

Data collection occurs once for each participant, with no intervention or follow-up required. Responses will remain anonymous, and no clinical procedures, biological samples, or physical assessments will be conducted. The study aims to generate foundational evidence that may inform future preventive strategies and wellness programs targeted at university students, particularly those in health-related fields.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years.
* Enrolled as an undergraduate Physical Therapy student.
* Able and willing to provide informed consent.

Exclusion Criteria:

* History of cardiovascular, metabolic, or psychiatric disorders.
* Current use of medications that affect appetite, sleep, or mood.
* Incomplete or inconsistent responses to the study questionnaires.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of undergraduate physical therapy students aged 18-30 years from various universities. This group represents a young adult population frequently exposed to high academic demands, lifestyle irregularities, and stress-related behaviors that may influence eating patterns, sleep quality, and early cardiovascular risk. Participants are generally healthy with no reported cardiovascular, metabolic, or psychiatric conditions.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Eating Attitudes Score (EAT-26) | 1 month, collected at baseline
  Total score on the Eating Attitudes Test (EAT-26) to assess disordered eating patterns and attitudes toward food. Higher scores indicate a greater risk of unhealthy eating behaviors.
Sleep Quality Score (PSQI) | 1 month, collected at baseline
  Global score from the Pittsburgh Sleep Quality Index (PSQI) evaluating sleep quality and disturbances. Higher scores reflect poorer sleep quality.
Perceived Stress Level (PSS-10) | 1 month, collected at baseline
  Description: Total score on the Perceived Stress Scale (PSS-10), measuring the degree to which participants perceive their lives as stressful. Higher scores indicate greater perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- EG Physio, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No